CLINICAL TRIAL: NCT01808703
Title: Clinical Trial of PeriZone PerioPatch in Subjects With Chronic Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MIS Implant Technologies, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PZ12-02; MIS Implant Technologies Ltd. (Other Grant/Funding Number: MIS Implant Technologies Ltd.)
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Periodontitis
Keywords: Periodontitis; Periodontal pocket; Periodontal diseases
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis; Periodontal Pocket; Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scaling and root planing plus PerioPatch (Experimental): All subjects in this group will receive scaling and root planing (full mouth during no more than 2 sessions within two weeks following the Baseline exam). Thereafter, PeriZone PerioPatch will be dispensed to subjects per randomization for administration over the trial period. Subjects will apply study patches (i.e., BID on Days 1, 28 and 42; QD on Days 2-6; Days 14-20, 29-30 and 43-44) to designated "treatment sites" (i.e., measuring 6 mm or more in pocket depth at Baseline).
  Interventions: Device: PeriZone PerioPatch; Procedure: Scaling and root planing alone
- Scaling and root planing alone (Active Comparator): Subjects in this group will receive only scaling and root planing (full mouth during no more than 2 sessions within two weeks following the Baseline exam).
  Interventions: Procedure: Scaling and root planing alone

INTERVENTIONS:
Device: PeriZone PerioPatch — The PeriZone PerioPatch is an approved barrier or device product intended for the management of all types of oral wounds, injuries and ulcerations of the gingival and oral mucosa (510K number K103054). PerioPatch devices will be applied adjunctively following scaling and root planing).
  Arms: Scaling and root planing plus PerioPatch
Procedure: Scaling and root planing alone — Following completion of the Baseline examination, all randomized patients will receive full mouth scaling and root planing at a maximum of two visits within a 14-day time period (Weeks -2 to 0). Use of hand curettes and/or ultrasonic instruments will be permitted. Local or topical anesthesia may be used for patient comfort at the discretion of the clinician performing the scaling and root planing.

SUMMARY:
The purpose of this study is to determine if a topical, adhesive patch (PeriZone PerioPatch) applied to the gums after a deep tooth cleaning (scaling and root planing) reduces the signs of advanced gum disease (chronic periodontitis) more than the deep tooth cleaning alone. Eighty patients with advanced gum disease will be recruited and treated within this clinical trial. Patients will be evaluated for changes in gum measurements over a 12-week period.

DETAILED DESCRIPTION:
Objectives: 1) to evaluate the efficacy of PeriZone PerioPatch (FDA approved device, 510K number K103054) in reducing pocket depth (PD) in subjects with moderate to severe chronic periodontitis; and 2) to assess the effect of PeriZone PerioPatch on secondary clinical outcomes associated with chronic periodontitis including bleeding on probing (BOP), clinical attachment level (CAL), Gingival Index (GI) and Plaque Index (PI).

Participants: A total of 80 participants with generalized moderate to severe chronic periodontitis will be recruited for this clinical trial.

Trial Design: This study is a multicenter, randomized, single blind, and controlled design trial with two parallel arms. The 2 arms of the study are:

* Arm A - Scaling and root planing plus PeriZone PerioPatch;
* Arm B - Scaling and root planing alone (control group).

Procedures (methods): After potential patients have been screened, informed consent forms are signed, and patients have completed the remaining screening evaluations, each patient will be randomized to a treatment group. Patients must present with generalized, moderate to severe chronic periodontitis defined as having at least two periodontal pockets measuring 6 mm or more and bleeding on probing (at Baseline).

Periodontal probing measurements (PD, CAL, GI and PI) will be performed at Baseline (prior to randomization), and at Weeks 4, 8 and 12. All subjects will receive scaling and root planing (full mouth during at most 2 sessions within two weeks following the Baseline exam). Thereafter, PeriZone PerioPatch will be dispensed to subjects per randomization for administration over the trial period (i.e., Days 1-6; Days 14-20; Days 28-30; Days 42-44). Intraoral soft tissue inspection will be performed at Screening, Baseline and at Weeks 4, 8 and 12. Adverse event collection will be performed at Weeks 4, 8 and 12. Compliance will be will be evaluated via collection of unused study devices.

Analysis Plan: Baseline and demographic data will be summarized by treatment. Adverse events and safety outcomes will be categorized by treatment and summarized with descriptive statistics. Changes in probing depths, bleeding scores, clinical attachment levels Gingival Index and Plaque Index scores (from Baseline) will be expressed as means per subjects and tested for inter-group differences using nonparametric rank analysis of covariance.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females 18 years or older
* Able and willing to follow study procedures and instructions
* Must have read, understood and signed an informed consent form
* Present with at least 12 teeth in the functional dentition, excluding third molars
* Generalized, moderate to severe chronic periodontitis
* Present with at least two periodontal pockets (on separate teeth) measuring 6 mm or more and that bleed on probing

Exclusion Criteria:

* Gross oral pathology
* Chronic treatment (i.e., two weeks or more) with anti-inflammatory medications (steroids or nonsteroidal anti-inflammatory drugs) or any other medications known to affect periodontal status (e.g., phenytoin, calcium antagonists, cyclosporine and coumadin) within one month of the screening examination
* Antibiotic treatment within 3 month prior to the screening examination
* History of rheumatic fever, valvular disease, valve replacement or prosthetic joint replacement necessitating antibiotic prophylaxis
* Active infectious diseases such as hepatitis, human immunodeficiency virus (HIV) or tuberculosis
* Reported allergies to herbal products
* Taking herbal product supplements
* Severe unrestored caries or any condition that is likely to require antibiotic treatment over the study
* Periodontal therapy (quadrant or maintenance scaling and root planing and/or periodontal surgical therapy) within 6 months prior to enrollment.
* Female patients who report being pregnant or lactating, or female patients who are of childbearing potential and who are not using hormonal, barrier methods of birth control (e.g., oral or parenteral contraceptives, diaphragm plus spermicide, condoms), or abstinence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Change in pocket depth (PD)from Baseline | At 4, 8 and 12 weeks
  PD will be measured from the free gingival margin to the base of the pocket and will be recorded in whole millimeters (mm). If a PD reading falls between two millimeter readings, the rule shall be to round down and the lower of the two readings will be recorded. All sites with PD of 5 mm or more will have two PD readings recorded (multiple-pass probing measurements) per examination time point. The average of the two PD readings will be the basis for deciding whether the site qualifies for treatment (average of two PD readings of 6 mm or more) at Baseline and the response to treatment (Weeks 4, 8 and 12).

SECONDARY OUTCOMES:
Change in clinical attachment level (CAL) from Baseline | At 4, 8 and 12 weeks
  CAL will be measured as the linear distance from the cemento-enamel junction (CEJ) to base of the pocket in mm. The examining clinician will measure CAL directly or indirectly (PD - recession). If a CAL reading falls between two millimeter readings, the rule shall be to round down and the lower of the two readings will be recorded.
Change in percent bleeding on probing (BOP) from Baseline | At 4, 8 and 12 weeks
  Presence or absence of bleeding to manual probing recorded as a dichotomous variable as follows: 0 - No bleeding within 10 seconds after probing; 1 -Bleeding within 10 seconds after probing.
Change in Gingival Index (GI) from Baseline | At 4, 8 and 12 weeks
  Degree of gingival inflammation recorded on an ordinal scale of 0-3 as follows (Loe & Silness, 1963): 0- Normal gingiva; 1 - Mild inflammation (slight change in color, slight edema); no bleeding on palpation (i.e., sulcular sweep); 2 - Moderate inflammation (redness, edema, glazing); bleeding on palpation (i.e., sulcular sweep); 3 - Severe inflammation (i.e., marked redness, edema); ulceration, tendency to spontaneous bleeding.
Change in Plaque Index (PI) from Baseline | At 4, 8 and 12 weeks
  Relative amount of supragingival plaque recorded on an ordinal scale of 0-3 as follows (Silness & Loe, 1964: 0 - No plaque in the gingival area; 1 - A film of plaque adhering to the free gingival margin and the adjacent tooth. The plaque may be recognized only by running a probe across the tooth surface; 2 - Moderate accumulation of soft deposits within the gingival pocket and on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye; 3 - Abundance of soft matter within the gingival pocket and/or on the gingival margin and the adjacent tooth surface.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca S Wilder, MS, Principal Investigator — University of North Carolina, Chapel Hill; Gayle B McCombs, MS, Principal Investigator — Old Dominion University
Locations (2):
- United States (2):
  - School of Dentistry, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - G. W. Hirschfeld School of Dental Hygiene, Old Dominion University, Norfolk, Virginia